CLINICAL TRIAL: NCT07222579
Title: A Multicenter Phase II Study of Subcutaneous Blinatumomab for Treatment of Adult Patients With CD19-Positive Mixed Phenotype Acute Leukemia (MPAL)
Brief Title: Subcutaneous Blinatumomab for Treatment of Adult Patients With CD19-Positive Mixed Phenotype Acute Leukemia (MPAL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Ashkan Emadi, MD PHD, Alexander Bland Osborn Endowed Chair and Distinguished Professor, West Virginia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2506170190
Record Dates: First submitted 2025-10-20; First posted 2025-10-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: CD19 Positive; Mixed Phenotype Acute Leukemia (MPAL)
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute | interventions — blinatumomab

STUDY DESIGN:
Intervention Model Description: * Cohort A: Participants with newly diagnosed CD19+ MPAL who are ≥ 75 years old or deemed unfit for intensive chemotherapy
  * Cohort B: Participants with CD19+ MPAL in first or second CR/CRh/CRi with detectable MRD ≥0.1%
  * Cohort C: Participants with morphologic R/R CD19+ MPAL
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Blinatumomab in Newly Diagnosed CD19+ MPAL, Age ≥ 75 or Unfit for Intensive Chemotherapy (Experimental): Cohort A: Evaluate the efficacy of SC-blinatumomab in treating newly diagnosed CD19+ MPAL in patients ≥ 75 years old or those deemed unfit for intensive chemotherapy.
  * Each cycle = 34 days (26-day treatment period + 8-day treatment free interval between day 27 and day 34).
  * Cycle 1 receives treatment daily during the first week and 3 times (TIW) weekly (M/W/F) during weeks 2-4.
  * In subsequent cycles, the treatment will be administered TIW during weeks 1-4.
  * All subjects will be hospitalized for days 1-12 of cycle 1.
  * Other treatment doses will be given as outpatients. Subjects will remain in the outpatient department for 1-6 hours after each dose is given.
  * Treatment will be given with ability to delay cycle initiation based on blood counts or general physical/neurological examination findings per clinical indication and institutional standard practice.
  Interventions: Drug: Subcutaneous Blinatumomab
- Blinatumomab use in CD19+ MPAL in first or second CR/CRh/CRi with detectable MRD ≥0.1% (Experimental): Cohort B: Assess the ability of SC-blinatumomab to achieve MRD-negative CR in patients with CD19+ MPAL in CR/CRh/CRi with persistent MRD positivity (≥ 0.1%) after at least one line of treatment.
  * Each cycle = 34 days (26-day treatment period + 8-day treatment free interval between day 27 and day 34).
  * Cycle 1 receives treatment daily during the first week and 3 times (TIW) weekly (M/W/F) during weeks 2-4.
  * In subsequent cycles, the treatment will be administered TIW during weeks 1-4.
  * All subjects will be hospitalized for days 1-12 of cycle 1.
  * Other treatment doses will be given as outpatients. Subjects will remain in the outpatient department for 1-6 hours after each dose is given.
  * Treatment will be given with ability to delay cycle initiation based on blood counts or general physical/neurological examination findings per clinical indication and institutional standard practice.
  Interventions: Drug: Subcutaneous Blinatumomab
- Blinatumomab use in Morphologic R/R CD19+ MPAL (Experimental): Cohort C: Determine the efficacy of SC-blinatumomab in inducing CR, CRh, or CRi in patients with morphologic relapsed or refractory CD19+ MPAL.
  * Each cycle = 34 days (26-day treatment period + 8-day treatment free interval between day 27 and day 34).
  * Cycle 1 receives treatment daily during the first week and 3 times (TIW) weekly (M/W/F) during weeks 2-4.
  * In subsequent cycles, the treatment will be administered TIW during weeks 1-4.
  * All subjects will be hospitalized for days 1-12 of cycle 1.
  * Other treatment doses will be given as outpatients. Subjects will remain in the outpatient department for 1-6 hours after each dose is given.
  * Treatment will be given with ability to delay cycle initiation based on blood counts or general physical/neurological examination findings per clinical indication and institutional standard practice.
  Interventions: Drug: Subcutaneous Blinatumomab

INTERVENTIONS:
Drug: Subcutaneous Blinatumomab — Blinatumomab will be administered as a subcutaneous (SC) injection.
  Other Names: Blincyto®

SUMMARY:
This is a multicenter, non-randomized, open-label, phase II study evaluating blinatumomab administered subcutaneously in adult subjects with CD19+ MPAL. This trial consists of three cohorts of patients with CD19-positive MPAL, categorized as follows: 1. Cohort A: Newly diagnosed CD19+ MPAL in untreated patients who are either ≥ 75 years of age or have at least one coexisting condition precluding intensive chemotherapy. 2. Cohort B: Patients with CD19+ MPAL who have achieved complete remission (CR, CRh, or CRi) following at least one line of treatment but have detectable measurable residual disease (MRD) at a level of ≥ 0.1%, assessed using an assay with a minimum sensitivity of 0.01%. 3. Cohort C: Patients with CD19+ MPAL with morphologic relapsed or refractory (R/R) disease following at least one prior line of treatment. The Primary Objectives for each cohort are for Cohort A: to evaluate the efficacy of SC-blinatumomab in treatment; for Cohort B: to assess the ability of SC-blinatumomab to achieve MRD-negative CR; for Cohort C: to determine the efficacy of SC-blinatumomab in inducing CR, CRh, or CRi in patients.

At specified time points, subjects will undergo the following procedures: collection of informed consent, medical history, demographics, ECOG performance, and physical exam including vital signs as well as neurological examination including examination of writing ability. Subjects will provide samples for complete blood count with differential and blood chemistry profile, have a bone marrow aspiration and biopsy and lumbar puncture will be performed per protocol or if clinically indicated, and/or ECG, Echocardiography, pulmonary function test will be performed only if medically indicated.

The subcutaneous treatment will be given in both the inpatient and outpatient setting. For an individual subject the length of participation includes up to a 3-week screening period, up to a 13-month treatment period, and a safety follow-up visit (30 days after the last dose of study treatment), and a follow-up period.

ELIGIBILITY:
* Inclusion Criteria:
* General Criteria for all three Cohorts

  * Subjects must have histologically or cytologically confirmed MPAL based on 2022 WHO criteria
  * Subjects who have undergone allo-HSCT are eligible if they are ≥ 4 weeks post stem cell infusion, have no evidence of GVHD > Grade 2, and are at least ≥ 1 week off of immunosuppressive therapy. Per FDA recommendation, patients should be off of calcineurin inhibitors (CNIs) for at least 4 weeks before receiving blinatumomab
  * Subjects with a CNS leukemia must be clinically stable (i.e., asymptomatic with no focal neurological signs and symptoms, or signs and symptoms unchanged over 4 weeks with no > grade 2 manifestations) with a flow cytometric clear CSF in the 2 weeks prior to day 1 of SC-blinatumomab administration.
  * Ability to understand and willingness to sign a written informed consent document
  * Agree to comply with the study requirements and agree to come to the clinic/hospital for required study visits
  * Subjects with hematologic malignancies are expected to have hematologic abnormalities at study entry
* Specific Criteria for Cohort A

  o Subjects should be ineligible for available induction therapy either if they are 75 years of age or older or if they have at least one of the following coexisting conditions precluding intensive chemotherapy: a history of CHF for which treatment is warranted or a report of EF ≤50% in the last 12 months, a history of chronic stable angina, a report of DLCO of ≤65% or FEV1 ≤65% in the last 12 months, ECOG performance status 3 or 4, Charlson comorbidity index (CCI) ≥3.
* Specific Criteria for Cohort B

  * CD19+ MPAL in CR/CRh/CRi after at least one line of treatment with MRD positivity at a level of ≥0.1% using an assay with a minimum sensitivity of 0.01%.
  * ECOG performance status ≤2
  * Subjects must have organ function as below:

    * Direct bilirubin ≤ 2.5 mg/dL
    * AST/ALT/Alkaline phosphatase ≤ 5 X institutional upper limit of normal
    * Serum creatinine ≤ 3 mg/dL
* Specific Criteria for Cohort C

  * Confirmed R/R CD19+ MPAL
  * Previous cytotoxic chemotherapy (except for hydroxyurea) must have been completed by 5 half-lives of the drug(s) prior to day 1 of SC-blinatumomab. Per FDA recommendation, patients should have recovered to no more than Grade 1 toxicities from prior chemotherapy.
  * ECOG performance status ≤2
  * Subjects must have organ function as below:

    * Direct bilirubin ≤ 2.5 mg/dL
    * AST/ALT/Alkaline phosphatase ≤ 5 X institutional upper limit of normal
    * Serum creatinine ≤ 3 mg/dL
* Exclusion Criteria:
* Criteria for all three Cohorts

  * Subjects receiving any other investigational agents, or concurrent chemotherapy, radiation therapy, or immunotherapy for cancer treatment not including corticosteroids or hydroxyurea
  * Active, uncontrolled infection; subjects with infection under active treatment and controlled with antimicrobials are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Cohort A - Overall Survival | Up to 3 years
  The Overall Survival (OS) is the time from treatment initiation to death from any cause.
Cohort B - Rate of Complete Remission (CR), Complete Remission with Partial Hematological Recovery (CRh), or Complete Remission with Incomplete Hematological Recovery (CRi) with Minimal Residual Disease (MRD) negativity | At completion of 2 cycles (each cycle is 34 days)
  The rate of achievement of complete remission (CR/CRh/CRi) with MRD-negativity (<0.01%) after the first two cycles of therapy with blinatumomab. CR: Bone marrow blasts <5%; absence of circulating blasts; absence of extramedullary disease; absolute neutrophil count (ANC) ≥1000/µL and platelets ≥100,000/µL; MRD+ or unknown. CR +CRh: Bone marrow blasts <5%; absence of circulating blasts; absence of extramedullary disease; ANC ≥500/µL AND platelet count ≥50,000/µL. CR +CRi: Bone marrow blasts <5%; absence of circulating blasts; absence of extramedullary disease; with residual thrombocytopenia (platelet count of <100,000/µL) OR residual neutropenia (ANC <1000/µL); not fulfilling criteria for CRh. MRD Negativity: No detectable cancer cells using sensitive tests, with less than 0.01% cancer cells. MRD positivity indicates a higher risk of relapse, while MRD negativity is linked to long-term remission and survival benefits.
Cohort C - Rate of Complete Remission (CR) or Complete Remission with Partial Hematological Recovery (CRh) | At completion of 2 cycles (each cycle is 34 days)
  The rate of achievement of complete remission (CR/CRh) after the first two cycles of therapy with blinatumomab.
  Complete Remission (CR): No detectable cancer cells in the bone marrow (less than 5% blast cells) and normal blood counts. CRh: No detectable cancer cells, with partial recovery of blood counts (ANC 500-1,000/µL, platelets 50,000-100,000/µL). The rate of achieving these states is calculated by the proportion of patients who reach CR/CRh within a set time. Higher rates of achievement indicate that a larger proportion of participants are responding positively to the treatment, with no detectable cancer cells in their bone marrow and recovery of blood counts.

SECONDARY OUTCOMES:
Cohort A - MRD-negative CR + CRh rate | At completion of 2 cycles (each cycle is 34 days)
  MRD-negative CR + CRh rate is the proportion of participants who achieve either Complete Remission (CR) or Complete Remission with Partial Hematological Recovery (CRh) and also have no detectable minimal residual disease (MRD) in bone marrow. Higher rates of MRD-negative CR + CRh indicate the treatment is highly effective in both inducing remission and reducing the risk of relapse.
Cohort A - Event-Free Survival (EFS) | Up to approximately 3 years
  Time from treatment initiation to the earliest occurrence of one of the following events:
  * Failure to achieve CR, CRh, or CRi after at least two cycles of SC-blinatumomab
  * Relapse after achieving CR, CRh, or CRi
  * Initiation of new leukemia-directed therapy due to persistent disease or progression
  * Death from any cause
Cohort A - Incidence and Severity of Adverse Events (AEs) | Up to approximately 1 year
  The number of AE Incidences including the severity of those events. The descriptions and grading scales found in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, published on November 27, 2017, will be utilized for AE reporting. The general guidelines for each grade are Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Life-threatening), Grade 5 (Death).
Cohort B - Overall Survival | Up to approximately 3 years
  The Overall Survival (OS)is the time from treatment initiation to death from any cause.
Cohort B - Rate of MRD-negativity (<0.01%) | At completion of 1 cycle (cycle is 34 days)
  The rate of MRD-negativity (<0.01%) within one cycle of SC-blinatumomab treatment. MRD negativity means that the number of cancer cells is below the threshold of 0.01%. A higher rate of MRD negativity suggests that the treatment is highly effective in eliminating cancer cells and reducing the risk of relapse.
Cohort B - Event-Free Survival (EFS) | Up to approximately 1 year
  Time from treatment initiation to the earliest occurrence of one of the following events:
  * Failure to achieve CR, CRh, or CRi after at least two cycles of SC-blinatumomab
  * Relapse after achieving CR, CRh, or CRi
  * Initiation of new leukemia-directed therapy due to persistent disease or progression
  * Death from any cause
Cohort B - Incidence and Severity of Adverse Events (AEs) | Up to approximately 1 year
  The number of AE Incidences including the severity of those events. The descriptions and grading scales found in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, published on November 27, 2017, will be utilized for AE reporting. The general guidelines for each grade are Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Life-threatening), Grade 5 (Death).
Cohort C - Overall Survival | Up to approximately 3 years
  The Overall Survival (OS)is the time from treatment initiation to death from any cause.
Cohort C - Event-Free Survival (EFS) | Up to approximately 1 year
  Time from treatment initiation to the earliest occurrence of one of the following events:
  * Failure to achieve CR, CRh, or CRi after at least two cycles of SC-blinatumomab
  * Relapse after achieving CR, CRh, or CRi
  * Initiation of new leukemia-directed therapy due to persistent disease or progression
  * Death from any cause
Cohort C - Incidence and Severity of Adverse Events (AEs) | Up to approximately 1 year
  The number of AE Incidences including the severity of those events. The descriptions and grading scales found in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, published on November 27, 2017, will be utilized for AE reporting. The general guidelines for each grade are Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Life-threatening), Grade 5 (Death).
Overall - Incidence and Severity of Adverse Events (AEs) | Up to approximately 1 year
  The number of AE Incidences including the severity of those events. The descriptions and grading scales found in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, published on November 27, 2017, will be utilized for AE reporting. The general guidelines for each grade are Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Life-threatening), Grade 5 (Death).

OTHER OUTCOMES:
Overall - Characterization of Antigen Expression | Up to 10 years
  Assess CD19, CD81, and CD21 expression (levels) in leukemic blasts through flow cytometry and/or immunohistochemical staining to evaluate potential biomarkers of treatment response and resistance. High expression levels may correlate with better treatment outcomes, while low or absent expression may indicate resistance.
Overall - Frequency of Cytogenetic Abnormalities Identified by Karyotyping and Fluorescence In Situ Hybridization (FISH) | Up to approximately 10 years
  Percentage of patients with identified cytogenetic abnormalities and will be correlated descriptively with clinical outcomes including treatment response, relapse, and overall survival. The frequency and pattern of disease-specific chromosomal abnormalities detected by conventional karyotyping and fluorescence in situ hybridization (FISH) in leukemic blasts.
Overall - Frequency of Somatic Mutations Identified by Next-Generation Sequencing (NGS) and Polymerase Chain Reaction (PCR) | Up to approximately 10 years
  Percentage of patients with specific genetic alterations and explored for associations with treatment response, relapse patterns, and disease progression. The frequency and spectrum of somatic mutations, gene fusions, or rearrangements detected using next-generation sequencing (NGS) and/or polymerase chain reaction (PCR) in leukemic cells.
Overall - Transplantation and Cellular Therapy Outcomes | Up to approximately 3 years
  The proportion of subjects proceeding to allogeneic hematopoietic stem cell transplantation (alloHSCT) after SC-blinatumomab treatment, assessing their post-transplant outcomes, relapse rates, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Emadi, MD, Principal Investigator — WVU Cancer Institute
Locations (1):
- West Virginia University Cancer Institute, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No